CLINICAL TRIAL: NCT07330726
Title: The Efficacy of a Transmucosal Lidocaine Patch on Postoperative Pain Following Mandibular Third Molar Extraction
Brief Title: Lidocaine Patch and Lower Third Molar
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Shaimaa Mohsen, associate professor, Fayoum University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 37
Record Dates: First submitted 2025-12-28; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Impacted Third Molar Tooth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lidocaine patch (Experimental)
  Interventions: Drug: Lidocaine patch
- placeboo patch (Placebo Comparator)
  Interventions: Drug: placebo patch

INTERVENTIONS:
Drug: Lidocaine patch — transmucosal lidocaine patch after third molar tooth removal
  Arms: lidocaine patch
Drug: placebo patch — transmucosal placebo patch after third molar tooth removal
  Arms: placeboo patch

SUMMARY:
* Completed medical and dental history will take for all patients and the position of the impacted teeth will evaluate by panoramic films. Patients will fully inform about the treatment procedures, follow-up examinations and complications of surgical procedures.
* Full thickness mucoperiosteal flap will be raised to expose sufficient bone on lateral and distal aspect of the impacted molar. Removal of bone will be done with stainless steel bur under Constant irrigation with normal saline while removing bone to prevent thermal necrosis.
* When necessary, sectioning of crown and roots will be performed with a fissure bur. After tooth extraction, the alveolus will be inspected, curetted, and irrigated with 0.9% sterile saline solution.
* Surgical removal of impacted mandibular third molar will be done,1% metformin gel or placebo gel in the socket following removal of the impacted third molar .
* The mucoperiosteal flap will be repositioned and sutured with 3-0 black silk suture.
* Control side : use transmucosal placebo patch
* Study side: use transmucosal lidocaine patch Postoperative care
* Postoperatively, the patients were instructed to apply ice bags 20 min/hour for the next 6 hours to the surgical side, eat soft cold diet by the aid of a straw and to avoid hot diet and fluid on the day of surgery.
* Sutures were removed after 7 days postoperatively.
* All the patients will be evaluated on the 1st, 3rd, and 7th postoperative days for pain, preoperative and postoperative mouth opening, and degree of postoperative swelling.

ELIGIBILITY:
Inclusion Criteria:

* • Age ≥18ys

  * no systemic disease
  * impacted mandibular third molar class II position B on Pell- Gregory classification

Exclusion Criteria:

* • history of metabolic or systemic diseases affecting bone or healing process,

  * local infection,
  * tobacco use,
  * oral contraceptive,
  * pregnancy and lactation
  * patients who had taken analgesics or anti-inflammatories for 1 week prior to enrollment in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 7 days postoperative
  Pain was assessed using a visual analogue scale (VAS) of 10 units in combination with a graphic rating scale. On the VAS, the left most end represented the absence of pain (score 0) and the right most end indicated the most severe pain (score 10).